CLINICAL TRIAL: NCT00486538
Title: An Open-Label, Phase 2 Study to Evaluate the Efficacy and Tolerability of ABT-869 in Subjects With Advanced Renal Cell Carcinoma (RCC) Who Have Previously Received Treatment With Sunitinib
Brief Title: Study of ABT-869 in Subjects With Advanced Renal Cell Carcinoma Who Have Previously Received Treatment With Sunitinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M06-882
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Advanced Renal Cell Carcinoma
MeSH Terms: interventions — linifanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): One oral dose daily
  Interventions: Drug: ABT-869

INTERVENTIONS:
Drug: ABT-869 — One oral dose daily.

SUMMARY:
This study is designed to determine the clinical efficacy and toxicity of ABT 869 in the treatment of subjects with advanced renal cell carcinoma who have previously received treatment with sunitinib.

ELIGIBILITY:
Inclusion Criteria

* Subject has undergone previous nephrectomy.
* Subject has received at least 2 cycles (12 weeks) of treatment with sunitinib for RCC and stopped therapy due to progressive disease within 100 days prior to screening.
* Subject has measurable disease, defined as at least 1 unidimensionally measurable lesion on a CT scan as defined by RECIST.
* ECOG Performance Score of 0-1.
* No history of another active cancer within the past 5 years.Life expectancy of at least 4 months.
* Willing to take adequate measures to prevent pregnancy.

Exclusion Criteria

* Subject has received anti-cancer therapy within 21 days or within a period defined by 5 half lives, whichever is shorter, prior to study drug administration.
* Subject has untreated brain or meningeal metastases.
* Subject has received a tyrosine kinase inhibitor (TKI) other than sunitinib or sorafenib.
* Prior use of Avastin is allowed.
* The subject is receiving therapeutic anticoagulation therapy.
* The subject has a history of/or currently exhibits clinically significant cancer related events of bleeding (e.g., hematuria, hemoptysis).
* The subject currently exhibits symptomatic or persistent, uncontrolled hypertension defined as diastolic blood pressure (BP) > 100 mmHg; or systolic blood pressure (BP) > 150 mmHg.
* The subject has a history of myocardial infarction within 6 months of Study Day 1.
* The subject has a documented left ventricular (LV) Ejection Fraction < 50%.
* The subject has known autoimmune disease with renal involvement (eg, Lupus).
* Female subjects who are pregnant or breast feeding.
* Subject is receiving anti-retroviral therapy for HIV.
* Subject has a clinically significant uncontrolled condition(s) including but not limited to:

  * active uncontrolled infection,
  * Class III or IV heart failure as defined by the New York Heart Association functional classification system,
  * unstable angina pectoris or cardiac arrhythmia,
  * history of adrenal insufficiency,
  * psychiatric illness/social situation that would limit compliance with study requirements;
  * Active, ulcerative colitis, Crohn's disease, celiadisease or any other conditions that interfere with absorption.
  * Subject has a medical condition, which in the opinion of the study investigator places them at an unacceptably high risk for toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-06; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | From randomization until patient death or alive at 2 years

SECONDARY OUTCOMES:
Progression-free rate | Week 16
Best response rate | From randomization until patient death or alive at 2 years
Time to tumor progression | From randomization until patient death or alive at 2 years
Progression free survival | Radiographic evaluation every month, clinical evaluation every 4 weeks
Overall Survival | Two-year follow-up post study

CONTACTS AND LOCATIONS:
Overall Officials: Justin L. Ricker, MD, Study Director — AbbVie
Locations (13):
- United States (12):
  - Site Reference ID/Investigator# 7193, Sacramento, California
  - Site Reference ID/Investigator# 5243, Washington D.C., District of Columbia
  - Site Reference ID/Investigator# 5384, Chicago, Illinois
  - Site Reference ID/Investigator# 11662, Boston, Massachusetts
  - Site Reference ID/Investigator# 11663, Boston, Massachusetts
  - Site Reference ID/Investigator# 5379, Boston, Massachusetts
  - Site Reference ID/Investigator# 5380, Lebanon, New Hampshire
  - Site Reference ID/Investigator# 5249, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 6278, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 6269, Pittsburgh, Pennsylvania
  - Site Reference ID/Investigator# 7300, Charleston, South Carolina
  - Site Reference ID/Investigator# 6796, Houston, Texas
- Site Reference ID/Investigator# 6566, Vancouver, Canada

REFERENCES:
- [Derived] Tannir NM, Wong YN, Kollmannsberger CK, Ernstoff MS, Perry DJ, Appleman LJ, Posadas EM, Cho D, Choueiri TK, Coates A, Gupta N, Pradhan R, Qian J, Chen J, Scappaticci FA, Ricker JL, Carlson DM, Michaelson MD. Phase 2 trial of linifanib (ABT-869) in patients with advanced renal cell cancer after sunitinib failure. Eur J Cancer. 2011 Dec;47(18):2706-14. doi: 10.1016/j.ejca.2011.09.002. Epub 2011 Nov 10. PMID 22078932